CLINICAL TRIAL: NCT07182929
Title: Radiographic Assessment of Deproteinized Porcine Versus Bovine Bone Mineral in Sinus Augmentation: A Retrospective Study
Brief Title: Radiographic Assessment of Deproteinized Porcine Versus Bovine Bone Mineral in Sinus Augmentation
Status: Completed | Type: Observational
Sponsor: Guoli Yang (Other)
Collaborators: The Dental Hospital of Zhejiang University School of Medicine (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Guoli Yang, Professor, The Dental Hospital of Zhejiang University School of Medicine
Organization: The Dental Hospital of Zhejiang University School of Medicine (Other)
Other Study IDs: 2024-153(R); 81901051, 82370991, 2022KY872 (Other: National Natural Science Foundation of China (NSFC); Zhejiang Provincial Department of Science and Technology)
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Sinus Floor Elevation; Sinus Floor Augmentation
Keywords: clinical research; Sinus Floor Augmentation; Cone-beam computed tomography; Bone Substitutes; Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DBBM: Patients in DBBM group receive 0.5g of DBBM (Bio-Oss®, 0.25-1.0 mm, Geistlich Pharma AG Co., Ltd, Wolhusen, Switzerland) during the sinus augmentation
  Interventions: Procedure: Lateral Sinus Floor Augmentation with Deproteinized Porcine Bone Mineral
- DPBM: Patients in DBBM group receive 0.5g of DBBM (Bio-Oss®, 0.25-1.0 mm, Geistlich Pharma AG Co., Ltd, Wolhusen, Switzerland) during the sinus augmentation

INTERVENTIONS:
Procedure: Lateral Sinus Floor Augmentation with Deproteinized Porcine Bone Mineral — Lateral Sinus Floor Augmentation Using Deproteinized Porcine Bone Mineral (DPBM, test) with Simultaneous Implant Placement and 6-Month CBCT Follow-Up
  Groups: DBBM

SUMMARY:
The goal of this retrospective study is to compare the radiographic outcomes of deproteinized porcine bone mineral (DPBM) and deproteinized bovine bone mineral (DBBM) following lateral sinus floor augmentation (LSFA) with simultaneous implant placement. The main questions it aims to answer are:

Does DPBM show greater graft resorption than DBBM at 6 months postoperatively? Do both materials achieve comparable bone quality and osseointegration outcomes despite differences in resorption rates?

This is a retrospective, single-center cohort study. Participants included 56 patients (56 sinuses) who underwent LSFA with either DPBM (test group, n=28) or DBBM (control group, n=28) and had complete cone-beam CT scans taken preoperatively, immediately postoperatively, and at 6 months post-surgery. Radiographic parameters such as bone height, augmentation volume, and bone texture features were analyzed to evaluate graft stability and new bone formation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years;
2. Single or multiple missing teeth in the posterior maxilla with a healing period of at least 3 months;
3. Complete baseline data and surgical records;
4. Underwent LSFA with simultaneous placement of a single implant, grafted exclusively with either DBBM (Bio-Oss®, 0.25-1.0 mm, Geistlich Pharma AG, Wolhusen, Switzerland) or DPBM (THE Graft®, 0.25-1.0 mm, Purgo Biologics, Seoul, Korea);
5. Available CBCT images obtained preoperatively (T0), immediately postoperatively (T1), and at 6 months postoperatively (T2);
6. RBH ≤6 mm shown by CBCT at T0 at the edentulous site;
7. No systemic disease, untreated periapical pathology or active periodontitis;
8. Provision of written informed consent for the implant surgery by the patient or their legal guardian.

Exclusion Criteria:

1. Uncontrolled systemic diseases or any bone-metabolism diseases;
2. Pregnancy or lactation;
3. Head and neck radiation therapy within the past 5 years;
4. acute and chronic inflammation in the maxillary sinus;
5. Additional vertical or horizontal bone augmentation procedures besides LSFA;
6. Use of graft materials other than the specified DBBM or DPBM, or use of composite grafts;
7. Heavy smoking (≥20 cigarettes/day), alcohol abuse, or history of substance abuse;
8. Placement of multiple implants in the same grafted site (excluded to avoid within-patient confounding).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received LSFA with simultaneous implant placement from June 2022 to June 2024 at the Stomatology Hospital, Zhejiang University School of Medicine, were screened for eligibility. All patients underwent preoperative clinical, radiographic examinations and laboratory tests. Eligible patients subsequently received LSFA performed by experienced implant surgeons following the standardized surgical protocol.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Apical Bone Height (ABH) | immediately postoperatively (T1), and 6 months postoperatively (T2)
  The vertical distance (mm) from the implant apex to the most apical point of the graft material
Bone Height (BH) | immediately postoperatively (T1), and 6 months postoperatively (T2)
  The vertical distance (mm) from the implant shoulder to the most apical point of the graft material. Site-specific measurements were denoted as buccal (bBH), palatal (pBH), mesial (mBH), and distal (dBH) bone heights
Endo-Sinus Bone Gain (ESBG) | immediately postoperatively (T1), and 6 months postoperatively (T2)
  The vertical distance of the augmented bone along the longitudinal axis of the implant, from the sinus floor to the most apical point of the graft
augmented volume (AV, mm³) | immediately postoperatively (T1), and 6 months postoperatively (T2)
  The augmented volume (AV, mm³) was measured at both T1 and T2 and was analyzed with the segmentation function of 3D Slicer 5.8.1

SECONDARY OUTCOMES:
Peri-Implant Bone Level (PBL) | immediately postoperatively (T1), and 6 months postoperatively (T2)
  The distance (mm) between the most coronal and the most apical levels of the implant-bone/graft contact interface. Site-specific measurements were denoted as buccal (bPBL), palatal (pPBL), mesial (mPBL), and distal (dPBL) peri-implant bone levels

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital, School of Stomatology, Zhejiang University., Hangzhou, Zhejiang 310000, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the retrospective nature of the study and ethical considerations related to patient privacy.

REFERENCES:
- [Background] Krennmair S, Postl L, Schwarze UY, Malek M, Stimmelmayr M, Krennmair G. Clinical, radiographic, and histological/histomorphometric analysis of maxillary sinus grafting with deproteinized porcine or bovine bone mineral: A randomized clinical trial. Clin Oral Implants Res. 2023 Nov;34(11):1230-1247. doi: 10.1111/clr.14164. Epub 2023 Aug 23. PMID 37610063
- [Background] Galindo-Moreno P, Abril-Garcia D, Carrillo-Galvez AB, Zurita F, Martin-Morales N, O'Valle F, Padial-Molina M. Maxillary sinus floor augmentation comparing bovine versus porcine bone xenografts mixed with autogenous bone graft. A split-mouth randomized controlled trial. Clin Oral Implants Res. 2022 May;33(5):524-536. doi: 10.1111/clr.13912. Epub 2022 Mar 3. PMID 35224778
- [Background] Lee JS, Shin HK, Yun JH, Cho KS. Randomized Clinical Trial of Maxillary Sinus Grafting using Deproteinized Porcine and Bovine Bone Mineral. Clin Implant Dent Relat Res. 2017 Feb;19(1):140-150. doi: 10.1111/cid.12430. Epub 2016 Jun 21. PMID 27324175
- [Background] Cassetta M, Perrotti V, Calasso S, Piattelli A, Sinjari B, Iezzi G. Bone formation in sinus augmentation procedures using autologous bone, porcine bone, and a 50 : 50 mixture: a human clinical and histological evaluation at 2 months. Clin Oral Implants Res. 2015 Oct;26(10):1180-4. doi: 10.1111/clr.12423. Epub 2014 May 26. PMID 24861978
- [Background] Pagliani L, Andersson P, Lanza M, Nappo A, Verrocchi D, Volpe S, Sennerby L. A collagenated porcine bone substitute for augmentation at Neoss implant sites: a prospective 1-year multicenter case series study with histology. Clin Implant Dent Relat Res. 2012 Oct;14(5):746-58. doi: 10.1111/j.1708-8208.2010.00314.x. Epub 2010 Oct 26. PMID 20977615
- [Background] Barone A, Ricci M, Covani U, Nannmark U, Azarmehr I, Calvo-Guirado JL. Maxillary sinus augmentation using prehydrated corticocancellous porcine bone: hystomorphometric evaluation after 6 months. Clin Implant Dent Relat Res. 2012 Jun;14(3):373-9. doi: 10.1111/j.1708-8208.2010.00274.x. Epub 2010 May 11. PMID 20491813
- [Background] Iezzi G, Degidi M, Piattelli A, Mangano C, Scarano A, Shibli JA, Perrotti V. Comparative histological results of different biomaterials used in sinus augmentation procedures: a human study at 6 months. Clin Oral Implants Res. 2012 Dec;23(12):1369-76. doi: 10.1111/j.1600-0501.2011.02308.x. Epub 2011 Nov 2. PMID 22092377
- [Background] Scarano A, Piattelli A, Perrotti V, Manzon L, Iezzi G. Maxillary sinus augmentation in humans using cortical porcine bone: a histological and histomorphometrical evaluation after 4 and 6 months. Clin Implant Dent Relat Res. 2011 Mar;13(1):13-8. doi: 10.1111/j.1708-8208.2009.00176.x. PMID 19438954
- [Background] Orsini G, Scarano A, Piattelli M, Piccirilli M, Caputi S, Piattelli A. Histologic and ultrastructural analysis of regenerated bone in maxillary sinus augmentation using a porcine bone-derived biomaterial. J Periodontol. 2006 Dec;77(12):1984-90. doi: 10.1902/jop.2006.060181. PMID 17209782